CLINICAL TRIAL: NCT03866642
Title: Two Year Follow up of Cadence Total Ankle Replacement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Cadence-2019
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Ankle Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cadence Total Ankle Replacment — Cadence Total Ankle prosthesis

SUMMARY:
Over the last decades, total ankle replacement (TAR) emerged as a reliable treatment option in end-stage ankle osteoarthritis (OA) while preserving motion and physiological load. The Cadence™ is a fourth-generation, two-component, fixed-bearing implant with minimal tibial and talar resection. It has been in clinical use since July 2016, the purpose of this study was to compare the clinical outcome and radiological outcomes of total ankle arthroplasty with use of the Cadence™ prosthesis at St. Michael's Hospital.

DETAILED DESCRIPTION:
Over the last decades, total ankle replacement (TAR) emerged as a reliable treatment option in end-stage ankle osteoarthritis (OA) while preserving motion and physiological load. The Cadence™ is a fourth-generation, two-component, fixed-bearing implant with minimal tibial and talar resection. It has been in clinical use since July 2016, the purpose of this study was to compare the clinical outcome and radiological outcomes of total ankle arthroplasty with use of the Cadence™ prosthesis at St. Michael's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Ankle arthritis treated with Cadence Total Ankle Replacement system

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage ankle arthritis requiring surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | Two Years

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided